CLINICAL TRIAL: NCT02383381
Title: Pre and Post-operative Rectus Muscle Insertion Site Changing Using Anterior Segment Optical Coherence Tomography in Strabismus Patients
Brief Title: Lateral Rectus Muscle and Anterior Segment Optical Coherence Tomography (AS-OCT)
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-05-026-005
Record Dates: First submitted 2015-02-24; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2014-02

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: lateral rectus recession — typical surgery for correcting intermittent exotropia

SUMMARY:
•Background and study aims : The investigators conducted this study to evaluate the movement of extraocular muscle after strabismus surgery with non-invasive tool called AS-OCT.

* Who can participate? patients who underwent typical lateral rectus recession surgery for correcting intermittent exotropia
* What does the study involve? Volunteers will attend a clinic for four visits over six months. They will undergo AS-OCT at every visits during follow up period. AS-OCT is non-invasive test to evaluate operation site. The test only requires their cooperation when they undergo AS-OCT.
* What are the possible benefits and risks of participating? This is non-invasive test for your postoperative follow up. Therefore, there will be no risks about this test.
* Where is the study run from? Samsung Medical Center
* When is the study starting and how long is it expected to run for? From Feb 2014 to Dec 2014

DETAILED DESCRIPTION:
The aim of this study is 1) to evaluate the reliability and accuracy of AS-OCT in the measurement of the lateral rectus (LR) insertion distance, 2)to investigate the longitudinal change of LR muscle insertion after strabismus surgery, and 3)to determine the effect of insertion movement on the angle of deviation after strabismus surgery. An AS-OCT scan of the LR muscle was performed every visits. Preoperative limbus-LR insertion distance was compared with intraoperative surgical caliper measurement of LR insertion using intraclass correlation coefficient analysis (ICC). Data on gender, age, degree of deviation (prism diopter), and spur-LR insertion distance using AS-OCT were collected at postoperative months 1,3 6.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent lateral rectus recession surgery for correcting intermittent exotropia

Exclusion Criteria:

* previous ocular surgery
* other ocular diseases except intermittent exotropia
* amblyopia

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 patients : 21 males and 9 females age: 9 to 60 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The change of limbus-muscle insertion distance measured with AS-OCT | baseline and 1.3.6 months

REFERENCES:
- [Background] Liu X, Wang F, Xiao Y, Ye X, Hou L. Measurement of the limbus-insertion distance in adult strabismus patients with anterior segment optical coherence tomography. Invest Ophthalmol Vis Sci. 2011 Oct 28;52(11):8370-3. doi: 10.1167/iovs.11-7752. PMID 21948556
- See also: basic information of intermittent exotropia including treatment — http://eyewiki.aao.org/Intermittent_Exotropia